CLINICAL TRIAL: NCT06297395
Title: Mid-Term Outcomes Of Subaxial Cervical Traumatic Injuries in Assiut University Trauma Center
Brief Title: Subaxial Cervical Traumatic Injuries
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Peter Philip Phily Ishaq, Resident, Assiut University
Other Study IDs: Cervical Traumatic Inj
Record Dates: First submitted 2024-02-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Cervical Injury Spine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess the mid-term outcomes of treating subaxial cervical traumatic injury cases admitted to the Trauma Unit of Assiut University Hospital.

DETAILED DESCRIPTION:
Injuries to the subaxial cervical spine can be bony, discoligamentous or a combination of both. Cervical spine trauma is common resulting from high energy trauma such as falling from height and motor vehicle accident . The subaxial cervical spine is a common site of cervical injury with more than 50 % of injuries being located between C5 and C7 MRI is superior to CT scans for evaluating the spinal cord, nerve roots, disc, and ligamentous structures in the cervical spine There are a couple of classification systems that have been devised The first is the Subaxial Injury Classification System (SLIC). This classification stratifies the type of fracture, the competency of the DLC, and the patient's neurologic status with numerical values to determine the course of treatment.

A second classification system is the AO Spine Subaxial Cervical Spine Injury Classification. The AO Spine SCICS classifies injuries based on 4 parameters: injury morphology, facet involvement, neurological status, and case-specific modifiers Patients with fractures deemed unstable or neurologic compromise should undergo decompression and stabilization. Intervention within 24 hours of injury leads to better improvement in ASIA scores .

Although we receive and treat a large number of patients with various subaxial cervical traumatic injuries in Assiut University Hospital each year, there is uncertainty about the midterm outcome of the treatment we provide.

In this study, The investigators will assess the mid-term outcomes of all patients with subaxial cervical traumatic injuries who complete a minimum one year follow up regardless of the neurological status or treatment type used.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting with subaxial cervical spine traumatic injuries with and without cervical cord injury who complete a minimum of one year follow up

Exclusion Criteria:

* Patients who refuse to participate in the study Patients with pathological fractures

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients fulfilling the inclusion criteria presenting to our hospital will be included in the study (Total coverage). Based on hospital records, we usually receive around 100 cases each year. We will also include all patients prospectively recorded in our data base starting from 11-01-2022. This data base includes 96 to date.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of improvement | Baseline
  Percentage of improvement in NDI (Arabic version) following conservative and surgical treatment during the follow up visits

SECONDARY OUTCOMES:
Patient Outcomes | Baseline
  AO Spine PROST
Complication | Baseline
  Mortality rate
rehabilitation | Baseline
  Improvement of neurological deficit by ASIA score
Complication | Baseline
  Incidence and rate of complications
rehabilitation | Baseline
  Return to work and activity of daily living.
Complication | Baseline
  Need for admission to the Intensive Care unit.
Complication | Baseline
  Post traumatic respiratory distress.
Complication | Baseline
  Fracture healing - pseudarthrosis - implant failure.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad El- Sharkawi, Prof, Study Director — Assiut University

REFERENCES:
- [Background] Stauffer ES. Subaxial injuries. Clin Orthop Relat Res. 1989 Feb;(239):30-9. PMID 2912631
- [Background] Feuchtbaum E, Buchowski J, Zebala L. Subaxial cervical spine trauma. Curr Rev Musculoskelet Med. 2016 Dec;9(4):496-504. doi: 10.1007/s12178-016-9377-0. PMID 27864669
- [Background] Aebi M. Surgical treatment of upper, middle and lower cervical injuries and non-unions by anterior procedures. Eur Spine J. 2010 Mar;19 Suppl 1(Suppl 1):S33-9. doi: 10.1007/s00586-009-1120-8. Epub 2009 Oct 14. PMID 19826842
- [Background] Pourtaheri S, Emami A, Sinha K, Faloon M, Hwang K, Shafa E, Holmes L Jr. The role of magnetic resonance imaging in acute cervical spine fractures. Spine J. 2014 Nov 1;14(11):2546-53. doi: 10.1016/j.spinee.2013.10.052. Epub 2013 Nov 22. PMID 24269913
- [Background] Vaccaro AR, Koerner JD, Radcliff KE, Oner FC, Reinhold M, Schnake KJ, Kandziora F, Fehlings MG, Dvorak MF, Aarabi B, Rajasekaran S, Schroeder GD, Kepler CK, Vialle LR. AOSpine subaxial cervical spine injury classification system. Eur Spine J. 2016 Jul;25(7):2173-84. doi: 10.1007/s00586-015-3831-3. Epub 2015 Feb 26. PMID 25716661
- [Background] Shaheen AA, Omar MT, Vernon H. Cross-cultural adaptation, reliability, and validity of the Arabic version of neck disability index in patients with neck pain. Spine (Phila Pa 1976). 2013 May 1;38(10):E609-15. doi: 10.1097/BRS.0b013e31828b2d09. PMID 23429690
- [Background] Sadiqi S, Oner FC. A disease-specific patient reported outcome instrument for spine trauma is developed, validated and available! Re: Andrzejowski et al. Measuring functional outcomes in major trauma: can we do better? Eur J Trauma Emerg Surg. 2023 Jun;49(3):1605-1606. doi: 10.1007/s00068-022-02167-8. Epub 2022 Nov 15. No abstract available. PMID 36378305